CLINICAL TRIAL: NCT03780686
Title: The Effect of Adding Dopamine Infusion to Noradrenaline Infusion Combined With Restrictive Hydration on Renal Function and Tissue Perfusion During Open Abdominal Surgeries
Brief Title: Dopamine and Norepinephrine Infusion With Restricted Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayman Anis Metry, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ASUH3206/17
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Renal Function Test, Urine Output, Lactate Level
Keywords: Restrictive hydration,; Dopamine,; Norepinephrine,; Serum lactate,; Standard hydration
MeSH Terms: interventions — Norepinephrine; Dopamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dopamine and norepinephrine infusion (Active Comparator): Infusion doppamine (2-5mcg/kg/min) and norepinephrine (3mcg/kg/h) with restricted fluid
  Interventions: Drug: Norepinephrine, dopamine
- Norepinephrine (Active Comparator): Infusion norepinephrine (3mcg/kg/h) with restricted fluid.
  Interventions: Drug: Norepinephrine, dopamine
- Standard fluid management (No Intervention): Standard fluid managements.

INTERVENTIONS:
Drug: Norepinephrine, dopamine — drugs to decrease bleeding
  Arms: Dopamine and norepinephrine infusion; Norepinephrine

SUMMARY:
This study was designed to assess the effect of adding dopamine infusion in addition to restrictive hydration combined with noradrenaline infusion on intraoperative serum lactate levels as an indicator for tissue hypo perfusion and renal function in comparison to restrictive hydration combined with noradrenaline infusion only and standard hydration during open abdominal surgeries.

DETAILED DESCRIPTION:
One hundred and twenty patients were randomly assigned into three groups (dopamine norepinephrine group, restrictive hydration group and liberal hydration group) undergoing open abdominal procedures (radical cystectomy and hemi colectomy). In Restrictive group (n=40): Ringer's solution was infused at a rate of 1 ml.kg.h-1 until the basic part of the surgery (tumor resection) is completed to be followed by 3 ml.kg.h-1 of Ringer's solution until the end of surgery. Noradrenaline infusion (0.07mcg.kg.min-1) was combined with fluids until the end of surgery. In Liberal group (n=40): the conventional fluid replacement was introduced according to maintenance, deficit for the first 3 hours (hours fasting x body weight) and 3rd space loss (estimated between 8-10 ml.kg.h-1).

The outcome to be assessed was serial measurements of serum lactate intraoperatively and immediate postoperatively as an index of tissue perfusion, in addition to blood pressure, heart rate and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with American Society of Anesthesiologists (ASA) physical status I or II
* Age range from 18-80 years scheduled to either radical cystectomy or hemicolectomy were contained in the study.

Exclusion Criteria:

* Patients with coagulopathies,
* Hepatic dysfunction (prothrombin ratio <50%),
* Renal dysfunction,
* Congestive heart failure (New York Heart Association scores ≥3),
* Contraindications for epidural analgesia (e.g. patient refusal, local infection or coagulopathy), and peripheral vascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-04-09 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Changes in serum lactate level | Before induction of anesthesia and up to 12 hours after.
  Serum lactate level in mmol/l
Changes in renal function test | Before induction of anesthesia and up to 12 hours after.
  Measuring creatinine level

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No